CLINICAL TRIAL: NCT01664793
Title: From Innovation to Solutions: Autodialers, Use of Early Autumn Physicals and Vaccination Assessment as a Vital Sign to Increase Childhood Influenza Vaccination in Diverse Settings
Brief Title: From Innovation to Solutions: Childhood Influenza Vaccination Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Richard Zimmerman, Professor, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1U01IP000321-01 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-08-14 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Influenza
Keywords: influenza; vaccination; strategies; children/adolescents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group Year 1 (Experimental): The 4 Pillars Immunization Toolkit along with donated vaccines for early season vaccination, staff education and support.
  Interventions: Behavioral: 4 Pillars Immunization Toolkit
- Control Group Year 1 (No Intervention): Control sites will not receive assistance with increasing influenza vaccination in Year 1, they will follow guidelines for usual care.

INTERVENTIONS:
Behavioral: 4 Pillars Immunization Toolkit — Pillar 1: Convenient Vaccination Services; Pillar 2: Patient notification about the importance of vaccination and availability of convenient services; Pillar 3: Enhanced Office Systems; Pillar 4: Motivation: Office immunization champion tracks progress towards a goal; Early delivery of donated vaccines for disadvantaged children, staff education, support of effort by research staff.
  Arms: Intervention Group Year 1

SUMMARY:
The purpose of this study is to increase childhood influenza vaccination rates using the FDA licensed influenza vaccines according to national guidelines in a randomized cluster trial in which primary care offices are randomized to intervention or control with the control group receiving the intervention in the second year.

DETAILED DESCRIPTION:
The investigators will conduct a stratified, randomized cluster trial of 20 diverse primary care practices to compare influenza vaccination rates in intervention and control sites. Intervention sites will use a package of newly developed and evidence-based techniques that will be tailored to their practice structure and culture, called the 4 Pillars Immunization Toolkit, in addition to receiving donated vaccine for early season vaccination. Control practices will not receive such assistance but will receive the intervention in the second year.

ELIGIBILITY:
Inclusion criteria:

For children: attendance at the selected health care center within the last year and age >/=6 months thru 18 years.

Exclusion Criteria:

For children: Severe egg allergy or allergy to influenza vaccine

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 87665 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zimmerman, MD, MPH, Principal Investigator — University of Pittsburgh, School of Medicine, Department of Family Medicine and Clinical Epidemiology; Chyongchiou Lin, PhD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, School of Medicine, Deparment of Family Medicine and Clinical Epidemiology, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Nowalk MP, Lin CJ, Hannibal K, Reis EC, Gallik G, Moehling KK, Huang HH, Allred NJ, Wolfson DH, Zimmerman RK. Increasing childhood influenza vaccination: a cluster randomized trial. Am J Prev Med. 2014 Oct;47(4):435-43. doi: 10.1016/j.amepre.2014.07.003. Epub 2014 Aug 8. PMID 25113138
- [Background] Zimmerman RK, Nowalk MP, Lin CJ, Hannibal K, Moehling KK, Huang HH, Matambanadzo A, Troy J, Allred NJ, Gallik G, Reis EC. Cluster randomized trial of a toolkit and early vaccine delivery to improve childhood influenza vaccination rates in primary care. Vaccine. 2014 Jun 17;32(29):3656-63. doi: 10.1016/j.vaccine.2014.04.057. Epub 2014 Apr 29. PMID 24793941

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Children who are active patients of 10 diverse pediatric and family medicine practices and who had at least one visit between 3/1/2011 and 2/29/2012 will serve as the Intervention group; n=49,039.
  Intervention sites will use the 4 Pillars toolkit along with early season vaccine to promote increases in childhood influenza vaccination.
- Control Group: Children who are active patients of 10 diverse pediatric and family medicine practices and who had at least one visit between 3/1/2011 and 2/29/2012 will serve as the control group; n=38,626. They will receive the 4 Pillars Toolkit and early season vaccine in Year 2.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 49039 | 38626
Completed | 49039 | 38626
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Children enrolled at family medicine practices and pediatric practices in the year preceding the intervention year for both intervention and control groups who were seen for a visit between 3/1/2010 and 2/28/2011.
Groups:
- Intervention Group: Children in 10 diverse pediatric and family medicine practices. Baseline group are active patients of the practices with a visit between 3/1/2010 and 2/28/2011.
- Control Group: Children in 10 diverse pediatric and family practices. Baseline group are active patients of the practices with a visit between 3/1/2010 and 2/28/2011.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 43293 | 38306 | 81599
Age, Continuous [Mean (Standard Deviation); unit: years] — To be eligible, the practice must have had a patient population of children under 19 years old.
  years | 7.3 (4.8) | 7.1 (5.2) | 7.2 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21560 | 18540 | 40100
  Male | 21733 | 19766 | 41499
Region of Enrollment [Number; unit: children at sites]
  United States | 43293 | 38306 | 81599

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome
Description: Influenza vaccination rates in each arm at the end of year 1
Time Frame: 3/1/2011-2/29/2012
Measure: Number; unit: participants vaccinated out of all
Groups:
- Intervention Group: Children seen in 10 diverse pediatric and family medicine practices between 3/1/2011 and 2/29/2012.
- Control Group: Children with a visit between 3/1/2011 and 2/29/2012 in 10 diverse pediatric and family practices.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 49039 | 38626
participants vaccinated out of all | 26432 | 19352
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Chi-square tests for comparisons of between-arm changes in vaccination rates from pre to post intervention

2. Secondary Outcome: Effectiveness Score
Description: Two staff members from each site were surveyed as to usefulness/effectiveness of a list of strategies recommended in the toolkit to increase vaccination rates. Values (range = 1-100 with 1 being not at all effective and 100 being highly effective) were averaged and used as an effectiveness score for each strategy. The average value for each site was combined with all sites and averaged for each strategy. (actual range = 20.6-90.7).
Time Frame: End of February 2012
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: 2 respondents in each of 10 diverse pediatric and family medicine practices.
- Control Group: This group did not rate effectiveness of the intervention.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 0
units on a scale | 75 (14) |

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Intervention Group; Control Group: Children in 10 diverse pediatric and family medicine practices seen between 8/1/2011 and 2/29/2012. We used the number of children who were vaccinated during intervention as the denominator for adverse events, because there is no other study-related risk for non-vaccinated children.
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/26432 | 0/19352
Other Adverse Events (participants affected / at risk) | 0/26432 | 0/19352

LIMITATIONS AND CAVEATS:
2 offices of 1 practice were randomized to each arm potentially causing carryover of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No